CLINICAL TRIAL: NCT00005026
Title: A Phase I Feasibility Trial of Carboplatin and Topotecan Followed by Carboplatin and Paclitaxel (Sequential Doublets) in Patients With Previously Untreated Epithelial Ovarian Carcinoma and Primary Peritoneal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Stage III or Stage IV Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067547; GOG-9906
Record Dates: First submitted 2000-04-06; First posted 2004-02-25 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2008-07

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Paclitaxel; Topotecan

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have stage III or stage IV ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of administering multiple courses of carboplatin and topotecan without excessive dose modification or course delay in patients with previously untreated ovarian epithelial or primary peritoneal carcinoma. II. Describe the response rate and progression-free interval in these patients with this treatment regimen. III. Determine pharmacokinetic and pharmacodynamic parameters related to the sequence of carboplatin and topotecan administration in these patients.

OUTLINE: Patients are assigned to one of three treatment regimens. Regimen I: Patients receive carboplatin IV over 30 minutes on day 1 followed by topotecan IV over 30 minutes on days 1-3. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Regimen II: Patients receive topotecan IV over 30 minutes on days 1-3 followed by carboplatin IV over 30 minutes on day 3. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Regimen III: Patients receive topotecan IV over 30 minutes on days 1-5 followed by carboplatin IV over 30 minutes on day 5. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment continues every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 1 month and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 15-80 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV ovarian epithelial or primary peritoneal carcinoma Prior surgery required within the past 12 weeks Either optimal (no greater than 1 cm residual disease) or suboptimal residual disease following initial surgery No ovarian epithelial tumors of low malignant potential (borderline tumor) The following histologic epithelial cell types are eligible: Serous adenocarcinoma Mucinous adenocarcinoma Clear cell adenocarcinoma Transitional cell carcinoma Adenocarcinoma not otherwise specified Endometrioid adenocarcinoma Undifferentiated carcinoma Mixed epithelial carcinoma Malignant Brenner tumor

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least lower limit of normal Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT and alkaline phosphatase no greater than 2.5 times ULN No acute hepatitis Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No unstable angina No myocardial infarction within past 6 months Abnormal cardiac conduction (e.g., bundle branch block, heart block) allowed if stable for past 6 months Other: No septicemia or severe infection No severe gastrointestinal bleeding No concurrent or prior invasive malignancies within past 5 years except nonmelanoma skin cancer No greater than grade 1 neuropathy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics Other: No prior cancer treatment that contraindicates study protocol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Bookman, MD, Study Chair — Fox Chase Cancer Center
Locations (47):
- United States (46):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Tampa Bay Cancer Consortium, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Bookman MA, McMeekin DS, Fracasso PM. Sequence dependence of hematologic toxicity using carboplatin and topotecan for primary therapy of advanced epithelial ovarian cancer: a phase I study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Nov;103(2):473-8. doi: 10.1016/j.ygyno.2006.03.014. Epub 2006 May 2. PMID 16631245